CLINICAL TRIAL: NCT03529162
Title: A Prospective Randomized Study Comparing Suture Anchor and Soft Tissue Pectoralis Major Tendon Techniques for Biceps Tenodesis
Brief Title: A Prospective Study Comparing Suture Anchor and Soft Tissue Pectoralis Major Tendon Techniques for Biceps Tenodesis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19, followed by PI leaving institution.
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Howard M Place, Department Chair, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 29091
Record Dates: First submitted 2018-04-23; First posted 2018-05-18 (Actual); Results first posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Bicep Tendinitis; Biceps; Tenosynovitis; Biceps Tendon Disorder
Keywords: Biceps Tendinitis; Subpectoral biceps tenodesis; Biceps tendon disorder
MeSH Terms: conditions — Tenosynovitis

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Suture Anchor Technique (SA) (Active Comparator): If randomized to this group, the patient will receive an open subpectoral long head of biceps tenodesis technique whereby the long head of biceps is re-attached to the humerus using an FDA-approved suture anchor (SA) device for the suture anchor technique. The device to be used will be the Mitek Super Quick Anchor.
  Interventions: Procedure: Long head of Biceps Tenodesis
- Pectoralis Major Technique (PMT) (Active Comparator): If randomized to this group, the patient will receive an open subpectoral long head of biceps tenodesis technique whereby the long head of biceps is re-attached by suturing the biceps tendon into the pectoralis major tendon.
  Interventions: Procedure: Long head of Biceps Tenodesis

INTERVENTIONS:
Procedure: Long head of Biceps Tenodesis — Patients will be randomized into two different groups to compare biceps tenodesis techniques

SUMMARY:
This is a prospective randomized controlled trial comparing two common techniques of long head of biceps tendon tenodesis in shoulder surgery. Numerous techniques of biceps tenodesis currently exist and are commonly performed. We will be comparing the tenodesis procedure using a suture anchor device versus a technique where the tendon is simply sutured to the pectoralis major tendon.

DETAILED DESCRIPTION:
Biceps tenodesis is a commonly performed procedure in shoulder surgery. In many cases, it is performed in conjunction with a rotator cuff repair. Currently, biceps tenodesis is performed in many different ways depending on surgeon preference. First, the location of the tenodesis can vary, as surgeons may prefer a suprapectoral or subpectoral tenodesis location. In addition, the tenodesis fixation technique can also vary, as surgeons have the option to use a screw or suture anchor to perform the tenodesis. There have been numerous studies comparing these various techniques, including suprapectoral versus subpectoral techniques and screw versus suture anchor techniques. None of these studies have been conclusive, and there continues to be controversy as to the best technique.

The current study will compare two techniques of subpectoral biceps tenodesis. Specifically, we will compare tenodesis using a suture anchor versus a technique where the tendon is simply sutured to the pectoralis major tendon. The latter technique has been previously described and published.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 100 years
* Able to provide written informed consent
* Has: (a) partial- or full-thickness rotator cuff tear verified by preoperative magnetic resonance imaging (MRI) and arthroscopy; (b) concomitant biceps lesions (LHBT partial tear>50%, SLAP type II lesion, pulley lesion, or subluxation/dislocation of LHBT) that were diagnosed arthroscopically with concomitant symptoms; and (c) arthroscopic rotator cuff repair.

Exclusion Criteria:

* Any medical illness that adversely impacts the patient's ability to complete the study procedures
* Isolated glenohumeral pathological conditions
* Any prior surgery on the same shoulder
* Complete rupture of the LHBT assessed by MRI or at time of procedure
* Incomplete repair of the rotator cuff

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Kim, MD, Principal Investigator — St. Louis University
Locations (3):
- United States (3):
  - Saint Louis University, St Louis, Missouri
  - SSM Health - Saint Louis University Hospital, St Louis, Missouri
  - SSM Health - St. Mary's Hospital, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abbot AE, Li X, Busconi BD. Arthroscopic treatment of concomitant superior labral anterior posterior (SLAP) lesions and rotator cuff tears in patients over the age of 45 years. Am J Sports Med. 2009 Jul;37(7):1358-62. doi: 10.1177/0363546509331940. Epub 2009 Apr 13. PMID 19364887
- [Background] Ahmed M, Young BT, Bledsoe G, Cutuk A, Kaar SG. Biomechanical comparison of long head of biceps tenodesis with interference screw and biceps sling soft tissue techniques. Arthroscopy. 2013 Jul;29(7):1157-63. doi: 10.1016/j.arthro.2013.04.001. Epub 2013 May 29. PMID 23725678
- [Background] Chen CH, Hsu KY, Chen WJ, Shih CH. Incidence and severity of biceps long head tendon lesion in patients with complete rotator cuff tears. J Trauma. 2005 Jun;58(6):1189-93. doi: 10.1097/01.ta.0000170052.84544.34. PMID 15995469
- [Background] Chung SW, Oh JH, Gong HS, Kim JY, Kim SH. Factors affecting rotator cuff healing after arthroscopic repair: osteoporosis as one of the independent risk factors. Am J Sports Med. 2011 Oct;39(10):2099-107. doi: 10.1177/0363546511415659. Epub 2011 Aug 3. PMID 21813440
- [Background] Golish SR, Caldwell PE 3rd, Miller MD, Singanamala N, Ranawat AS, Treme G, Pearson SE, Costic R, Sekiya JK. Interference screw versus suture anchor fixation for subpectoral tenodesis of the proximal biceps tendon: a cadaveric study. Arthroscopy. 2008 Oct;24(10):1103-8. doi: 10.1016/j.arthro.2008.05.005. Epub 2008 Jun 16. PMID 19028161
- [Background] Habermeyer P, Magosch P, Pritsch M, Scheibel MT, Lichtenberg S. Anterosuperior impingement of the shoulder as a result of pulley lesions: a prospective arthroscopic study. J Shoulder Elbow Surg. 2004 Jan-Feb;13(1):5-12. doi: 10.1016/j.jse.2003.09.013. PMID 14735066
- [Background] Hsu AR, Ghodadra NS, Provencher MT, Lewis PB, Bach BR. Biceps tenotomy versus tenodesis: a review of clinical outcomes and biomechanical results. J Shoulder Elbow Surg. 2011 Mar;20(2):326-32. doi: 10.1016/j.jse.2010.08.019. Epub 2010 Nov 4. PMID 21051241
- [Background] Koh KH, Ahn JH, Kim SM, Yoo JC. Treatment of biceps tendon lesions in the setting of rotator cuff tears: prospective cohort study of tenotomy versus tenodesis. Am J Sports Med. 2010 Aug;38(8):1584-90. doi: 10.1177/0363546510364053. Epub 2010 Jun 15. PMID 20551285
- [Background] Oh JH, Kim SH, Ji HM, Jo KH, Bin SW, Gong HS. Prognostic factors affecting anatomic outcome of rotator cuff repair and correlation with functional outcome. Arthroscopy. 2009 Jan;25(1):30-9. doi: 10.1016/j.arthro.2008.08.010. Epub 2008 Oct 10. PMID 19111216
- [Background] Oh JH, Lee YH, Kim SH, Park JS, Seo HJ, Kim W, Park HB. Comparison of Treatments for Superior Labrum-Biceps Complex Lesions With Concomitant Rotator Cuff Repair: A Prospective, Randomized, Comparative Analysis of Debridement, Biceps Tenotomy, and Biceps Tenodesis. Arthroscopy. 2016 Jun;32(6):958-67. doi: 10.1016/j.arthro.2015.11.036. Epub 2016 Feb 23. PMID 26921128
- [Background] Park JS, Kim SH, Jung HJ, Lee YH, Oh JH. A Prospective Randomized Study Comparing the Interference Screw and Suture Anchor Techniques for Biceps Tenodesis. Am J Sports Med. 2017 Feb;45(2):440-448. doi: 10.1177/0363546516667577. Epub 2016 Oct 22. PMID 28146397
- [Background] Pogorzelski J, Horan MP, Hussain ZB, Vap A, Fritz EM, Millett PJ. Subpectoral Biceps Tenodesis for Treatment of Isolated Type II SLAP Lesions in a Young and Active Population. Arthroscopy. 2018 Feb;34(2):371-376. doi: 10.1016/j.arthro.2017.07.021. Epub 2017 Sep 9. PMID 28899638
- [Background] Ramos CH, Coelho JC. Biomechanical evaluation of the long head of the biceps brachii tendon fixed by three techniques: a sheep model. Rev Bras Ortop. 2016 Dec 30;52(1):52-60. doi: 10.1016/j.rboe.2016.12.008. eCollection 2017 Jan-Feb. PMID 28194382
- [Background] Scheibel M, Schroder RJ, Chen J, Bartsch M. Arthroscopic soft tissue tenodesis versus bony fixation anchor tenodesis of the long head of the biceps tendon. Am J Sports Med. 2011 May;39(5):1046-52. doi: 10.1177/0363546510390777. Epub 2011 Jan 21. PMID 21257843
- [Background] Walch G, Edwards TB, Boulahia A, Nove-Josserand L, Neyton L, Szabo I. Arthroscopic tenotomy of the long head of the biceps in the treatment of rotator cuff tears: clinical and radiographic results of 307 cases. J Shoulder Elbow Surg. 2005 May-Jun;14(3):238-46. doi: 10.1016/j.jse.2004.07.008. PMID 15889020
- [Background] Zehnder Sw, Kaar SG, Joy E. Transpectoral Biceps Sling Tenodesis: Surgical Technique. Tech Should Surg. 2011;12: 32-35.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pectoralis Major Technique (PMT) | Suture Anchor Technique (SA)
Started | 2 | 2
Completed | 0 | 0
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Suture Anchor Technique (SA) | Pectoralis Major Technique (PMT) | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Median (Full Range); unit: years] | 51 [41 to 61] | 43 [41 to 45] | 47 [41 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
The American Shoulder and Elbow Surgeons Shoulder Score (ASES) [Median (Full Range); unit: scores on a scale] — The American Shoulder and Elbow Surgeons Shoulder Score (ASES) is a mixed outcome reporting measure, applicable for use in all patients with shoulder pathology regardless of their specific diagnosis.
  The ASES score contains a physician-rated and patient-rated section; however, only the pain visual analog scale (VAS) and 10 functional questions are typically used to tabulate the reported ASES score. The total score - 100 maximum points - is weighted 50% for pain and 50% for function. A score of 100 represents a better outcome and a score of 0 represents a worse outcome.
  scores on a scale | 23.3 [6.67 to 40] | 25.0 [15 to 35] | 25 [6.67 to 40]
The Disabilities of the Arm, Shoulder and Hand Score (DASH) [Median (Full Range); unit: scores on a scale] — The disabilities of the arm, shoulder and hand (DASH) questionnaire is a self-administered region-specific outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms. The DASH consists mainly of a 30-item disability/symptom scale, scored 0 (no disability) to 100.
  scores on a scale | 49.5 [45 to 54] | 62 [32 to 92] | 49.5 [32 to 92]
Visual Analog Scale (VAS) [Median (Full Range); unit: score on a scale] — The Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be'. The patient is asked to mark their pain level on the line between the two endpoints. "0" is no pain and "10" is pain as bad as it could be on the scale. The score on a scale represents the number, or score, that the patient selected to for their level of pain.
  score on a scale | 8.5 [7 to 10] | 9 [8 to 10] | 9 [7 to 10]
Single Assessment Numeric Evaluation (SANE) [Median (Full Range); unit: score on a scale] — The Single Assessment Numeric Evaluation (SANE) is a simple, one-question patient-reported outcome measure (PROM). Scoring is 1 to 100, with 100 being the highest function/no pain score.
  score on a scale | 35 [30 to 40] | 12.5 [0 to 25] | 27.5 [0 to 40]
Long Head of the Biceps Tendon Score (LHB) [Median (Full Range); unit: scores on a scale] — The LHB score is a composite endpoint (maximum 100 points) that evaluates 'biceps pain and muscle cramps', 'cosmesis', and 'flexion strength at the elbow'. It is an outcome score specific for biceps tendon pathology. The score range is 0-100, with a higher score representing better outcome. Population: Baseline data was not collected on one subject for this measure and the patient was lost to follow up for subsequent scoring.
  scores on a scale
    number analyzed (Participants) | 1 | 2 | 3
    (all) | 80 [80 to 80] | 38 [34 to 42] | 42 [34 to 80]

OUTCOME MEASURES:

1. Primary Outcome: Change in Long Head of the Biceps Tendon Score (LHB)
Description: The LHB score is a composite endpoint (maximum 100 points) that evaluates 'biceps pain and muscle cramps', 'cosmesis', and 'flexion strength at the elbow'. It is an outcome score specific for biceps tendon pathology. The score range is 0-100, with a higher score representing better function. The values represent the scores at 3 and 6 months, not a change of values from Baseline to 3 and 6 months.
Time Frame: This score obtained pre-operatively, and post-operatively at 3 months, 6 months, which are reported.
Population: Sample size too small. Baseline data was collected on three of the four subjects and due to COVID-19 and the PI leaving research institution, additional long-term data not collected on remaining subjects.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Pectoralis Major Technique (PMT) | Suture Anchor Technique (SA)
Number analyzed (Participants) | 2 | 1
units on a scale
  3 Month Data | 57.5 [30 to 85] | 89 [89 to 89]
  6 Month Data: number analyzed (Participants) | 0 | 1
  6 Month Data |  | 94 [94 to 94]

2. Secondary Outcome: Change in Visual Analogue Scale (VAS)
Description: The Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be'. The patient is asked to mark his pain level on the line between the two endpoints. "0" is no pain and "10" is the worst pain. The values represent the scores at 3 and 6 months, not a change of values from Baseline to 3 and 6 months.
Time Frame: This score obtained pre-operatively, and post-operatively at 3 months, 6 months, which are reported.
Population: Sample size too small. Baseline data was collected on all four subjects, but due to COVID-19 and the PI leaving research institution, additional long-term data not collected on all subjects. One subject was lost to follow up for outcome measure time frames.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Suture Anchor Technique (SA) | Pectoralis Major Technique (PMT)
Number analyzed (Participants) | 1 | 2
score on a scale
  3 Month Data | 3 [3 to 3] | 5.50 [2 to 9]
  6 Month Data: number analyzed (Participants) | 1 | 0
  6 Month Data | 2 [2 to 2] |

3. Secondary Outcome: Change in Disabilities of the Arm, Shoulder, and Hand Score (DASH)
Description: The disabilities of the arm, shoulder and hand (DASH) questionnaire is a self-administered region-specific outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms. The DASH consists mainly of a 30-item disability/symptom scale, scored 0 (no disability) to 100. The values represent the scores at 3 and 6 months, not a change of values from Baseline to 3 and 6 months.
Time Frame: This score obtained pre-operatively, and post-operatively at 3 months, 6 months, which are reported.
Population: as for outcome 2
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Suture Anchor Technique (SA) | Pectoralis Major Technique (PMT)
Number analyzed (Participants) | 1 | 2
score on a scale
  3 Month Data | 28 [28 to 28] | 51 [6 to 96]
  6 Month Data: number analyzed (Participants) | 1 | 0
  6 Month Data | 10 [10 to 10] |

4. Secondary Outcome: Change in Single Assessment Numeric Evaluation (SANE)
Description: The Single Assessment Numeric Evaluation (SANE) is a simple, one-question patient-reported outcome measure (PROM). Scoring is 1 to 100, with 100 being the highest function/no pain score. The values represent the scores at 3 and 6 months, not a change of values from Baseline to 3 and 6 months.
Time Frame: This score obtained pre-operatively, and post-operatively at 3 months, 6 months, which are reported.
Population: as for outcome 2
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Suture Anchor Technique (SA) | Pectoralis Major Technique (PMT)
Number analyzed (Participants) | 1 | 2
units on a scale
  3 Month Data | 50 [50 to 50] | 52.5 [7 to 98]
  6 Month Data: number analyzed (Participants) | 1 | 0
  6 Month Data | 70 [70 to 70] |

5. Secondary Outcome: Change in American Shoulder and Elbow Surgeons (ASES) Shoulder Score
Description: The American Shoulder and Elbow Surgeons Shoulder Score (ASES) is a mixed outcome reporting measure, applicable for use in all patients with shoulder pathology regardless of their specific diagnosis.
  The ASES score contains a physician-rated and patient-rated section; however, only the pain visual analog scale (VAS) and 10 functional questions are typically used to tabulate the reported ASES score. The total score - 100 maximum points - is weighted 50% for pain and 50% for function. A score of 100 represents a better outcome and a score of 0 represents a worse outcome. The values represent the scores at 3 and 6 months, not a change of values from Baseline to 3 and 6 months.
Time Frame: This score obtained pre-operatively, and post-operatively at 3 months, 6 months, which are reported.
Population: as for outcome 2
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Suture Anchor Technique (SA) | Pectoralis Major Technique (PMT)
Number analyzed (Participants) | 1 | 2
score on a scale
  3 Month Data | 65 [65 to 65] | 49.2 [16.7 to 81.7]
  6 Month Data: number analyzed (Participants) | 1 | 0
  6 Month Data | 78.3 [78.3 to 78.3] |

ADVERSE EVENTS:
Time Frame: Adverse event data was reviewed at each study visit during course of study. Six months was the maximum that patients were followed.
Description: No adverse events were reported in the four subjects.
Arm/Group | Suture Anchor Technique (SA) | Pectoralis Major Technique (PMT)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

LIMITATIONS AND CAVEATS:
Early termination of study due to COVID-19 and later the departure of PI from institution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-05): https://cdn.clinicaltrials.gov/large-docs/62/NCT03529162/Prot_SAP_002.pdf
  • Informed Consent Form (2019-03-19): https://cdn.clinicaltrials.gov/large-docs/62/NCT03529162/ICF_003.pdf